CLINICAL TRIAL: NCT05490797
Title: Effects of Mobile Application Dexteria Fine Motor Skills on Hand Dexterity and Grip Strength in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0255
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Ischemic; Skill, Social; Occlusion
Keywords: Stroke, Ischemic; Skill, Social; Occlusion
MeSH Terms: conditions — Ischemic Stroke; Social Skills; Bites and Stings

STUDY DESIGN:
Intervention Model Description: total 22 participants will be enrolled. In experimental group app based training will be performed along with conventional hand fine motor skills and dexterity therapy. Conventional hand therapy will be given to the second group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- app based training with conventional therapy (Experimental): In experimental group app based training will be performed along with conventional hand fine motor skills and dexterity therapy.
  Interventions: Other: app based training with conventional therapy
- conventional therapy (Active Comparator): The control group will receive conventional hand function rehabilitation therapy including, strengthening exercises which consist of palm down wrist flexion exercise, dexterity( shifting exercise) and fine motor skills(nine peg hole exercise)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: app based training with conventional therapy — The experimental group will receive an additional mobile application therapy including , dexterity fine motor skills, bowling game, scribble game and peglight game in addition to the conventional therapy for hand function.
  Arms: app based training with conventional therapy
Other: conventional therapy — conventional hand function rehabilitation therapy including, strengthening exercises which consist of palm down wrist flexion exercise, dexterity( shifting exercise) and fine motor skills(nine peg hole exercise)
  Arms: conventional therapy

SUMMARY:
To determine the effects of mobile application dexteria fine motor skills on hand dexterity and grip strength in chronic stroke patients

DETAILED DESCRIPTION:
This study will be conducted to investigate the effects of mobile applications of dexterity fine motor skills on hand dexterity and grip strength in chronic stroke patients. Data will be collected from Jinnah hospital Lahore and Riphah Rehabilitation center Lahore. All 22 patients will be taken using random sampling. Both study groups will be given common treatment of conventional hand function. The subjects will randomly assign to the experiment group with mobile apps training and the control group without mobile app training. Mobile applications like Dexteria, ScribbleKid, PegLight and Bowling game will be used for the purpose of training and success rate will be considered as outcome measure. Test and tools include the Nine Hole Peg Test (NHPT), the Fugl-Meyer Motor assessment (FMA), The Box & Block Test (BBT), and Grip strength will be assessed using a hand dynamometer. SPSS 25 version will be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Six months to 2 years post stroke
* Participants must be able to open and close their fingers (even only 2 cm of movement)
* Before stroke there must be fully functional hand
* Normal or intact vision

Exclusion Criteria:

* Neurological disorders other than stroke for example multiple sclerosis or Parkinson disease.
* Upper extremities acute orthopaedic conditions.
* Any cardiopulmonary complications
* Medically unstable patients.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
The Nine Hole Peg Test (NHPT) | 9 months
  The Nine Hole Peg Test (NHPT) is designed to quantify finger dexterity with neurological diagnoses patients.
Fugl-Meyer Motor assessment (FMA) | 9 months
  Fugl-Meyer Motor assessment (FMA) is specific for post stroke performance based on impairment index. This is specific for quantification of balance and motor functioning.
The Box &Block Test (BBT) | 9 months
  The Box &Block Test (BBT) is designed for measuring overall manual dexterity.
hand dynamometer. | 9 months
  Grip strength is assessed using a hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lanas F, Seron P. Facing the stroke burden worldwide. Lancet Glob Health. 2021 Mar;9(3):e235-e236. doi: 10.1016/S2214-109X(20)30520-9. Epub 2021 Jan 7. No abstract available. PMID 33422188
- [Background] Doumas I, Everard G, Dehem S, Lejeune T. Serious games for upper limb rehabilitation after stroke: a meta-analysis. J Neuroeng Rehabil. 2021 Jun 15;18(1):100. doi: 10.1186/s12984-021-00889-1. PMID 34130713
- [Background] Olsen TS. Arm and leg paresis as outcome predictors in stroke rehabilitation. Stroke. 1990 Feb;21(2):247-51. doi: 10.1161/01.str.21.2.247. PMID 2305400
- [Background] Jensen M, Thomalla G. Causes and Secondary Prevention of Acute Ischemic Stroke in Adults. Hamostaseologie. 2020 Feb;40(1):22-30. doi: 10.1055/s-0039-1700502. Epub 2019 Oct 24. PMID 31648355